CLINICAL TRIAL: NCT07351032
Title: Neural Mechanism of Skill Transfer in Parkinson's Disease
Brief Title: Understanding How Movements Are Transferred From Task to Task in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Caroline Paquette, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 24-12-053
Record Dates: First submitted 2025-09-26; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: PARKINSON DISEASE (Disorder)
Keywords: Transcranial Magnetic Stimulation; Split-belt Treadmill; Gait; Motor Adaptation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active rTMS First followed by Sham rTMS Second (Other): Session 1: active rTMS (iTBS) over the right PPC Session 2: sham rTMS (iTBS) over the right PPC
  Interventions: Other: Transcranial Magnetic Stimulation Active; Other: Transcranial Magnetic Stimulation Sham
- Sham rTMS First followed by Active rTMS Second (Other): Session 1: sham rTMS (iTBS) over the right PPC Session 2: active rTMS (iTBS) over the right PPC
  Interventions: Other: Transcranial Magnetic Stimulation Active; Other: Transcranial Magnetic Stimulation Sham

INTERVENTIONS:
Other: Transcranial Magnetic Stimulation Active — ACTIVE: intermittent Theta Burst Stimulation (a patterned form of rTMS). The participants will receive iTBS (50hz bursts at 5Hz for 600 pulses for a total duration of 3-minutes) over the right PPC at 80% RMT of the FDI.
Other: Transcranial Magnetic Stimulation Sham — SHAM: 2 coils on top of each other will be used instead of 1. The coil furthest to the head will be reversed. The coil on the head will not be stimulating but the reversed coil will (current directed away from the brain) with stimulate with the same parameters at the active stimulation (intermittent Theta Burst Stimulation (a patterned form of rTMS). The participants will receive iTBS (50hz bursts at 5Hz for 600 pulses for a total duration of 3-minutes) over the right PPC at 80% RMT of the FDI.

SUMMARY:
The purpose of this study is to understand how a specific brain area, the Posterior Parietal Cortex (PPC), plays a role in movement transfer from walking on a split-belt treadmill (SBT) to walking on the ground in people with Parkinson's disease (PwPD).

Here, investigators will apply repeated transcranial magnetic stimulation (rTMS) to upregulate the PPC. Then, the differences in the gait parameters between pre- and post-interventions will be compared between the TMS-active and the TMS-sham.

DETAILED DESCRIPTION:
The split-belt training has been shown to modulate gait in PwPD, but the skill transfer from the SBT training to the overground walking is poorly understood.

In this project, the subjects will visit the lab on three occasions: day 1 is for the clinical assessment based on the questionnaires, the 10-Meter Walk Task, as well as finding TMS targets and thresholds for the tibialis anterior (TA) and first dorsal interosseous (FDI) muscles, day 2 and day 3 are for either rTMS-active or rTMS-sham intervention. The second and third visits will take place at least 48h a part to ensure that the rTMS effects are washed out between visits.

During these two visits, the participants will first perform pre-overground walking tests (3 minutes): straight walking, steering, and turning, followed by pre-SBT adaptation tests (4 minutes) where they will adapt their gait to the asymmetrical belt that changes every 30 seconds. After these walking tests, the threshold measured on the first day will be validated, and the cortical excitability of the PPC will be measured by using a dual-coil: one is over the TA hotspot, and the other is over the PPC. Then, rTMS or sham intervention will be performed, followed by measuring the cortical excitability of the PPC. Immediately after that intervention, the participants will train on the SBT for 30 minutes in total (with a one-minute break every 5 minutes) with the speed of the belt changing every 30 seconds. Following the SBT training, the participants will perform post-overground and post-SBT adaptation tests. Lastly, the cortical excitability of the PPC will be measured.

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of idiopathic Parkinson's disease
* absence of freezing of gait confirmed by a "No" answer to the second item of the New Freezing of Gait Questionnaire (NFOGQ) and no observation of FOG during a freezing provoking test
* no other neurological diagnosis
* no severe musculoskeletal/orthopedic or vestibular condition that interferes with walking and or significantly affects balance
* no mild cognitive impairment (Montreal Cognitive Assessment ≥ 25)
* able to walk independently and without assistive device for 30 minutes
* no previous experience with split-belt treadmill.

Exclusion Criteria:

* severe dyskinesia that interacts with walking and balance hearing or visual impairment
* observed inability to walk safely on a tied-belt treadmill
* neurological disorders other than PD or other pathology (e.g., orthopedic) interfering with mobility. - contradiction for TMS
* implanted deep brain stimulator.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Stride length | Day 2 and Day 3
  The forward distance travelled by a foot during a gait cycle (cm) measured during overground walking and on the SBT with the Ambulatory Parkinson's Disease Monitoring (APDM) mobility lab system.
  A higher score indicates better gait control.
Dual Support | Day 2 and Day 3
  The percentage of the gait cycle when both feet are in contact with the ground (%) will be measured during overground walking and on the SBT with the Ambulatory Parkinson's Disease Monitoring (APDM) mobility lab system.
  A higher score indicates a longer time for both feet to be in contact with the ground.

SECONDARY OUTCOMES:
Cadence | Day 2 and Day 3
  The number of steps per minute will be measured during overground walking and on the SBT with the Ambulatory Parkinson's Disease Monitoring (APDM) mobility lab system.
  A higher score indicates better gait control.
Gait Speed | Day 2 and Day 3
  The speed of the subject, measured as the distance traveled in the gait cycle divided by the gait cycle duration (m/s) during overground walking and on the SBT will be measured with the Ambulatory Parkinson's Disease Monitoring (APDM) mobility lab system.
  A higher score indicates better gait control.
Turning Velocity | Day 2 and Day 3
  The peak angular velocity of the turn (deg/s) during overground walking will be measured with the Ambulatory Parkinson's Disease Monitoring (APDM) mobility lab system.
  The higher score indicates better turning performance.
Steps in turn | Day 2 and Day 3
  The number of steps taken in one turn during overground walking will be measured with the Ambulatory Parkinson's Disease Monitoring (APDM) mobility lab system.
  The higher score indicates better turning performance.
Step length | Day 2 and Day 3
  The distance between the heels of two consecutive steps (m) during overground walking will be measured with a custom MATLAB script.
  The higher score indicates better gait control.
Cortical Excitability | Day 2 and Day 3
  The cortical excitability will be assessed using a dual coil setup where two coils are placed on 2 different locations of the scalp at the same time. One coil will be positioned over the PPC, and the other over the TA hotspot.
  A total of 50 stimuli will be randomly delivered: 25 pulses will be applied solely over the TA hotspot (TA), and the other 25 paired pulses in which a PPC stimulus precedes the TA stimulus by 4 milliseconds (PPC + TA).
  Cortical excitability will be quantified by using the following ratio: (PPC + TA) / (TA).
  The higher score indicates the greater excitability of the neurons along the PPC-M1 pathway.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Paquette, PhD, Principal Investigator — McGill University
Locations (1):
- McGill University - Currie Gymnasium, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
We have a data management plan in place but will make anonymized data available.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT07351032/Prot_SAP_000.pdf